CLINICAL TRIAL: NCT04542616
Title: Outcomes Comparison Between Baerveldt 350 and Ahmed ClearPath 250 Tube Shunts for the Treatment of Glaucoma
Brief Title: Baerveldt 350 vs Ahmed ClearPath 250 for the Treatment of Glaucoma
Acronym: B350vsCP250
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Asher Weiner, MD, Clinical Associate Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00004680
Record Dates: First submitted 2020-08-27; First posted 2020-09-09 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Glaucoma
Keywords: Glaucoma; Baerveldt 350; Ahmed ClearPath 250
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: Comparison between 2 groups of patients requiring tube shunt implantation to treat their severe uncontrolled glaucoma. One group will receive a unilateral Baerveldt 350 tube shunt and the other a unilateral Ahmed ClearPath 250 tube shunt. The patients will be sequentially randomized into one of these tube shunts.
Who Masked: Outcomes Assessor
Masking Description: All patients will sign a consent form indicating they will be randomly receiving one of the 2 tube shunt models. It would be impossible to mask the patient or care provider to the type of tube shunt a patient received. The patients cannot bias the clinical data recorded on their follow up exams. All data will be recorded objectively. The outcome assessor will be masked to the type of shunt used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Baerveldt 350 (Active Comparator): The patients in this arm will receive a Baerveldt 350 tube shunt implantation for the treatment of their severe uncontrolled glaucoma.
  Interventions: Device: Baerveldt 350 vs. Ahmed ClearPath 250 tube shunt implantation
- Ahmed ClearPath 250 (Active Comparator): The patients in this arm will receive an Ahmed ClearPath 250 tube shunt implantation for the treatment of their severe uncontrolled glaucoma.
  Interventions: Device: Baerveldt 350 vs. Ahmed ClearPath 250 tube shunt implantation

INTERVENTIONS:
Device: Baerveldt 350 vs. Ahmed ClearPath 250 tube shunt implantation — Baerveldt 350 vs. Ahmed ClearPath 250 tube shunt implantation for the treatment of severe uncontrolled glaucoma.

SUMMARY:
To compare the safety and efficacy of Baerveldt 350 and Ahmed ClearPath 250 tube shunts in lowering IOP in glaucoma patients.

DETAILED DESCRIPTION:
Tube shunt implantation is a common type of surgery considered standard of care for treating significant potentially-blinding glaucoma where medical and laser treatment, and previous surgeries, have failed to control intra-ocular pressure (IOP) sufficiently to stop glaucoma progression towards blindness.

Since a larger plate tube (e.g., Baerveldt 350) is more difficult to implant requiring longer surgical time and intraoperative ocular muscle manipulation with possible patient discomfort, a smaller plate tube shunt (e.g., Ahmed ClearPath 250) requiring shorter surgical time and no ocular muscle manipulation may have an advantage if the long term surgical outcomes were the same.

However, the literature is lacking regarding the effect of the tube plate size on the final outcomes of tube shunt implantation. Most published comparisons are between totally different types of tube shunts regardless of plate size, often made of different materials, often comparing valved vs. non-valved tube shunts,combining different plate sizes in the same study groups,5 mixing tubes with or without combined cataract surgery in the same study groups, or comparing surgeries performed by several surgeons utilizing different surgical methods. Further, all these studies utilize tubes implanted into the anterior chamber (AC) thus increasing the risk of corneal failure, with no comparisons at all between tube shunts implanted through the ciliary sulcus of the eye designed to reduce the risk of corneal failure. Our Principle Investigator (AW) is specializing and well-published in this type of tube shunt implantation.

This prospective randomized trial is designed to resolve all these confusing factors in the literature and finally provide the answer of whether tube plate size has an effect on the final outcomes of tube shunt implantation by performing a "clean" study that would isolate the effect of tube plate size on long term outcomes. To achieve this goal our study will utilize two non-valved tube shunts with a different plate size (350 vs. 250 mm2) made of identical materials, in eyes that have already had cataract surgery, and all performed by the same surgeon (AW) through the ciliary sulcus.

ELIGIBILITY:
Inclusion Criteria:

* Significant uncontrolled glaucoma despite medical, laser or previous surgical therapy that requires tube shunt implantation as standard-of-care to stabilize the glaucoma and preserve vision.
* Pseudophakia
* Patients who are willing to participate and are able to understand and sign the study consent form.
* Age ≥18 years.

Exclusion Criteria:

* Phakic eyes (no previous cataract surgery).
* Aphakic eyes (status post previous cataract removal but without a lens implant).
* Age <18 years.
* Women of child-bearing age.
* Patients unable to comprehend and sign the study consent form.
* Women who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in intraocular pressure | 2 years
  Change in Intraocular pressure between preoperative baseline and postoperative follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Asher Weiner, MD, Principal Investigator — The Ross Eye Institute
Locations (1):
- The Ira G. Ross Eye Institute, Buffalo, New York, United States